CLINICAL TRIAL: NCT03809884
Title: Diet or Additional Supplement to Increase Potassium Intake: An Adaptive Clinical Trial
Brief Title: Dietary Counseling or Potassium Supplement to Increase Potassium Intake in Patients With High Blood Pressure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20180873-01H
Record Dates: First submitted 2018-12-13; First posted 2019-01-18 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
Keywords: High blood pressure; Potassium; Potassium Citrate; Dietary Counselling; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Potassium Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Counselling (Experimental): All enrolled patients will undergo a 1:1 counselling with a registered dietitian (with possible inclusion of family members, as appropriate). The dietitian will undertake an assessment of the comorbidities (e.g. diabetes), dietary intake, dietary habits (e.g. eating out, food preparation, socio-cultural aspects) and provide an individually tailored strategy to increase potassium in the diet. Secondly, on a weekly basis, the dietitian will contact the patient by telephone, or electronically (as preferred by the patient) to reinforce the advice and provide support/advice as necessary.
  Interventions: Behavioral: Dietary Counselling
- Potassium Citrate Supplement (Active Comparator): Patients who are not able to successfully increase their potassium intake at 4 weeks with dietary counselling will receive potassium citrate supplements. They will receive oral potassium supplementation in the form of 50 to 100 mmol of potassium citrate (as 25 to 50 ml of the liquid solution).
  Interventions: Behavioral: Dietary Counselling; Drug: Potassium Citrate

INTERVENTIONS:
Behavioral: Dietary Counselling — Individually tailored strategy to increase potassium in the diet.
Drug: Potassium Citrate — Dosing of 50 to 100 mmol of potassium citrate per day (as 25 to 50 ml of the liquid solution).
  Other Names: K-Citra
  Arms: Potassium Citrate Supplement

SUMMARY:
High blood pressure is the leading cause of cardiovascular disease worldwide. Many medicines are available to lower blood pressures successfully, as well as many non-medical options, such as dietary changes. Some effective dietary changes include decreasing sodium and increasing potassium in the diet. A lot of focus has been on sodium intake yet; potassium intake in the diet remains low amongst adult Canadians. Excellent data exist in the published research reporting that increasing potassium intake, either as diet or even as supplements, reduces blood pressure and reduces risk of cardiovascular outcomes such as stroke.

The overall purpose of this study is to reveal the most effective way of increasing potassium, amongst participants with high blood pressure whose existing intake of potassium is low. In the first stage, participants with high blood pressure and proven low potassium intake will receive dietary counselling. If after 4 weeks, there has not been a desired increase in potassium intake, the patients will be prescribed an additional potassium supplement.

DETAILED DESCRIPTION:
High blood pressure is the leading cause of cardiovascular disease worldwide, including in Canada. The prevalence of high blood pressure is steadily rising, with growing and ageing population. Many medicines are available to decrease blood pressures successfully, as well as many non-medical options, such as dietary changes and exercise. There is a marked preference amongst patients, reiterated in a recent Hypertension Canada report, for more research into methods for controlling blood pressure without medicines or to reduce the burden of taking many pills to control high blood pressure. Indeed, effective options do exist, especially with diet, specifically decreasing sodium and increasing potassium in diet. Both these recommendations are also made by organizations worldwide including the World Health Organization as well as Hypertension Canada. Though a lot of focus has been on sodium intake in the public health outreach, even the potassium intake in diet remains woefully low amongst adult Canadians. Excellent data exist in the published research reporting that increasing potassium intake, either as diet or even as supplements, reduces blood pressure and reduces risk of cardiovascular outcomes such as stroke. The advice most often provided is to 'eat more fruits and vegetables' which does not get translated into concrete change.

The Investigators propose to do a clinical trial in two stages (as an adaptive trial design). In the first stage, participants with high blood pressure and proven low potassium intake (measured on the basis of collecting urine for 24 hours) will get individually tailored dietary advice, reinforced by weekly supportive phone/email support. If at 4 weeks, there has not been a desired increase in potassium intake, the patients will be prescribed an additional potassium supplement. Testing at 4 weeks will be conducted again to confirm the efficacy of the potassium supplement. Final measurements will be planned at 52 weeks to observe and measure the persistence of the effect of diet or additional supplement. Concurrent measurements of sodium intake, blood pressure, participant satisfaction, safety measures will also be done.

The results of the study would help determine the most effective method of increasing potassium intake, thus reducing blood pressure, need for blood pressure lowering medicines, at the same time potentially increasing participant satisfaction. The current guidelines recommend changes in diet (not supplement) to increase potassium intake, hence the two stage design will only add supplements if the most rigorous dietary advice does not work. The Investigators have received letters of support from the World Hypertension League and Hypertension Canada in support of the research design and for dissemination and implementation of the findings.

ELIGIBILITY:
Inclusion Criteria:

1. Provides signed and dated informed consent form
2. Diagnosis of hypertension (either on treatment; or not on treatment with an ambulatory blood pressure monitor (ABPM)- daytime systolic blood pressure (SBP) > 140 or diastolic blood pressure (DBP) > 90)
3. Male or female, aged 18 and greater (women of child bearing potential must use highly effective contraception (e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants; intrauterine device (IUD) or intrauterine system (IUS); vasectomy of male partner and tubal ligation)
4. 24-Hour Urine K < 60 mmol/day

Exclusion Criteria:

1. Serum Potassium < 3.3 or > 5.1 mmol/L
2. Glomerular Filtration Rate < 45 ml/min/1.73m2
3. Primary hyperaldosteronism
4. Pregnancy or lactation
5. Psychiatric disorder which, in the opinion of the investigator, would interfere with the study, or inability to give consent
6. Severe Liver disease
7. Metabolic Alkalosis (HCO3 > 32 mmol/L)
8. Exclude patients who need to be started on renin-angiotensin-aldosterone blockade in the first 3 months
9. Gastrointestinal disorder (e.g. delayed gastric emptying, dysphagia, oesophageal/gastric/duodenal ulcer)
10. Presence of cardiac disease (sever myocardial damage, heart failure, or clinical changes in congestive heart failure, ejection fraction <35%)
11. Uncontrolled diabetes mellitus (HbA1C >12%)
12. Acute dehydration
13. Extensive tissue damage (burns)
14. Increased hypersensitivity to potassium (e.g. paramyotonia congenital or adynamia episodica hereditaria)
15. Patients taking other potassium supplements for another indication (eg. kidney stones)
16. Acidosis (pH<7.11)
17. Adrenal insufficiency
18. Allergies to any of the investigational product ingredients (medicinal and non- medicinal)
19. Patients on any of the following medications should be on a stable dose: angiotensin converting enzyme (ACE) inhibitors, angiotensin II receptor blockers, beta-blockers, mineralocorticoid receptor antagonists, amiloride, non steroidal antiinflammatory drugs (NSAIDs), beta-blockers, digoxin, and heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Successful increase in potassium intake | 4 weeks
  As estimated by 24 hour urine results at 4 weeks, achieving a urinary sodium > 90 mmol/day.

SECONDARY OUTCOMES:
Persistence of increase in potassium intake at 52 weeks | 52 weeks
  As estimated by comparison of persistence of change in potassium intake (as estimated by 24 hour urine results) from 4 weeks to 52 weeks.
Hyperkalemia Events | 4 weeks to 52 weeks
  Any episodes of hyperkalemia (as defined as a serum potassium greater than the 5.1 mmol/L)
Gastrointestinal Events | 4 weeks to 52 weeks
  Gastrointestinal side effects, specifically changes in bowel habits, belching and/or flatulence; abdominal pain or cramps.

CONTACTS AND LOCATIONS:
Overall Officials: Swapnil Hiremath, MD MPH, Principal Investigator — The Ottawa Hospital
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hiremath S, Fergusson D, Knoll G, Ramsay T, Kong J, Ruzicka M. Diet or additional supplement to increase potassium intake: protocol for an adaptive clinical trial. Trials. 2022 Feb 14;23(1):147. doi: 10.1186/s13063-022-06071-9. PMID 35164833